CLINICAL TRIAL: NCT05115513
Title: Examine the Feasibility of a Standardized Field Test for Marijuana Impairment: Laboratory Evaluations II
Brief Title: Standardized Field Test for Marijuana Impairment II
Acronym: NHTSA-II
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Highway Traffic Safety Administration (NHTSA) (U.S. Federal Agency); Hartford Hospital (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Godfrey Pearlson, Professor of Psychiatry and Neuroscience, Founding Director Olin Neuropsychiatry Research Center, Yale University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HHC-2021-0333; DTNH2216C00022 (Other: Department of Transportation); 2000032628 (Other: Yale IRB)
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Marijuana Impairment
Keywords: Marijuana; THC; Cannabis; Driving; Impairment; Intoxication
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Marijuana (Experimental): Placebo Marijuana will be administered.
  Interventions: Drug: Placebo THC
- Medium THC Marijuana (Experimental): Medium THC marijuana will be administered.
  Interventions: Drug: Medium THC

INTERVENTIONS:
Drug: Medium THC — Marijuana flower with medium THC
  Arms: Medium THC Marijuana
Drug: Placebo THC — Marijuana flower with no THC
  Arms: Placebo Marijuana

SUMMARY:
This research responds to NHTSA's request with a proposal to increase our understanding of smoked cannabis' (CNB's) acute effects on driving-relevant cognition and simulated driving performance, the persistence of these deficits over the hours after use, and the influence of prior experience with CNB on these effects. This extension study will aim to further investigate marijuana impaired behavior, using a similar design to our previous NHTSA Examine the Feasibility of a Standardized Field Test for Marijuana Impairment and the prior NIDA Neuroscience of Marijuana-Impaired Driving award, that used similar techniques and measures to quantify marijuana impaired automobile driving. We will be utilizing tasks and assessments that were shown to be strong indicators for cognitive and driving impairment in our NHTSA study.

DETAILED DESCRIPTION:
The proposed study was based upon a careful and thorough review of the scientific literature describing CNB effects on cognitive test performance and driving, as well as current state-of-knowledge on the sensitivity of biological assays for identifying recent CNB use. The study will carefully characterize the persistence of CNB's acute effects on cognitive test performance and driving over a several-hour time span. This will allow us to identify the point at which any effects of CNB intoxication driving-related cognitive tests, and driving performance cannot be distinguished from normal, i.e., the first step towards establishing standards for legal and social policy. The data obtained from simulated driving, cognitive tests, and biological assays of THC will be used in analyses aimed at identifying what tests or combination of tests predict both recent use and driving impairment risk.

This study will consist of 2 days (screening visit and dose visit). In a non-randomized, single blinded study, we will dose participants with placebo and high THC marijuana, about an hour apart, using paced inhalation through a vaporizer, an efficient means of delivering a standard THC dose. Participants will be told that the order they receive the doses will be random but they will always receive the placebo first, followed by the high dose. This will allow for standardization across all subjects and comparative values between placebo and drug. After inhaling the placebo dose, participants will be asked to complete one round of cognitive testing and a shortened version of the driving simulator (10 mins vs 30 mins). Approximately one hour post placebo dose, subjects will be administered high THC marijuana. Following this dosing, we will assess impairment through cognitive testing as well as a simulated driving test and neuropsychological tests. Samples of blood will also be collected at multiple time points throughout the study visits to be measured for THC concentration and its metabolites. This allows clarification between the relationship of impairment, as well as subjective and objective intoxication, and levels of THC and it's metabolites in the users system.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 yrs/ old
* Current driver's license and history of repeated highway vehicle driving experience (at least 2 years)
* Recent, recurrent CNB use and felt high when used
* Able to read, speak, and understand English
* Able and willing to provide written informed consent, and willing to commit to the study protocol

Exclusion Criteria:

* Current marijuana tolerance, desire to cut down, or cravings to use during periods of abstinence
* New CNB users who have not used at least once during their lifetime.
* Positive screen for drug and alcohol (except THC) on test day will result in rescheduling the appointment
* Former CNB users who are abstaining
* Pregnancy, breastfeeding, and ineffective birth control methods.
* History of adverse psychological or medical effects following cannabis use
* serious medical, neuro-ophthalmological, or neurological illness (i.e. cancer, seizure disorders, encephalopathy)
* History of head trauma with loss of consciousness > 30 minutes or concussion lasting 30 days.
* IQ <80 on the Wechsler Abbreviated Scale of Intelligence
* Inability to comprehend written instructions using the WRAT 4 reading achievement test
* Any medical/neurological condition that could compromise neurocognitive performance (i.e. epilepsy, multiple sclerosis, fetal alcohol syndrome)
* Uncontrolled, persistent high blood pressure
* Anyone deemed unsafe to study personnel for any reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Marijuana induced performance changes on Cogstate Groton Maze Learning task. | Post placebo at 30 minutes and post active dose administration at: 30 minutes, 60 minutes , 90 minutes, 120 minutes, 150 minutes, 180 minutes.
  The Cogstate Groton Maze Learning task assesses spatial learning and memory, it will be administered prior to dosing and at various time points after dosing.
Marijuana induced performance changes on Inquisit Maze Learning task. | Post placebo at 30 minutes and post active dose administration at: 30 minutes, 60 minutes , 90 minutes, 120 minutes, 150 minutes, 180 minutes.
  The Inquisit Maze Learning task assesses spatial learning and memory, it will be administered prior to dosing and at various time points after dosing.
Marijuana induced performance changes on the Time Reproduction Task. | Post placebo at 30 minutes and post active dose administration at: 30 minutes, 60 minutes , 90 minutes, 120 minutes, 150 minutes, 180 minutes.
  The Time Reproduction Task assesses general motor coordination plus timing, it will be administered prior to dosing and at various time points after dosing.

SECONDARY OUTCOMES:
Change in concentration of THC/metabolites in blood samples. | Post placebo at 5 minutes and post active dose administration at: 30 minutes, 60 minutes , 90 minutes, 120 minutes, 150 minutes, 180 minutes.
  Blood samples with be collected at 5 times throughout each day to assess for changes of THC and its metabolite levels.
Change in performance on simulated driving Road Tracking Task. | Post placebo at 10 minutes and post active dose administration at 210 minutes.
  The Road Tracking Task measures operational control of the vehicle. Operational control is measured by standard deviation of lane position from the center point of the lane.

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey Pearlson, M.D, Principal Investigator — Yale University
Locations (1):
- Olin Neuropsychiatry Research Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No